CLINICAL TRIAL: NCT04967014
Title: A Randomized, Open-label, Multiple-Dose, Crossover Phase 1 Clinical Trial to Evaluate the Safety and Pharmacodynamic/Pharmacokinetic Characteristics After Oral Administration of HIP2101 in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Safety and Pharmacodynamic/Pharmacokinetic Characteristics of HIP2101 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ESOL-101
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: Healthy Adult Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period I : RLD2104 Period II : HIP2104
  Interventions: Drug: HIP2101; Drug: RLD2101
- Sequence B (Experimental): Period I : HIP2104 Period II : RLD2104
  Interventions: Drug: HIP2101; Drug: RLD2101

INTERVENTIONS:
Drug: HIP2101 — Test drug
Drug: RLD2101 — Reference drug

SUMMARY:
A Phase 1 Study to Evaluate the Safety and Pharmacodynamic/Pharmacokinetic Characteristics of HIP2101 in Healthy Volunteers

DETAILED DESCRIPTION:
A Randomized, Open-label, Multiple-dose, Crossover Phase 1 Clinical Trial to Evaluate the Safety and Pharmacodynamic/Pharmacokinetic Characteristics after Oral Administration of HIP2101 in Healthy Adult Volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers in the age between 19 and 50 years old.
* Body mass index (BMI) in the range of 18 to 30 kg/m2 and weight 50.0kg to 90.0kg.
* After fully hearing and understanding the details of this clinical trial, Subjects who have willingness to sign of informed consent before the screening.
* Subject who are eligible from physical examination, clinical laboratory test by investigators judgment.

Exclusion Criteria:

* Gastrointestinal disorders (Crohn's disease or Acute/chronic pancreatitis) or gastrointestinal surgery (except for simple cecal or hernia surgery) which may affect the safety and pharmacokinetic evaluation of test drug.
* Subjects who have a history of hypersensitivity or clinically significant hypersensitivity to investigational product or the same component or other drugs.
* Aspartate aminotransferase and alanine aminotransferase exceed 2 times the upper limit of normal range from screening laboratory results before randomization.
* Subject who continues to drink (21 units / week, 1 unit = 10 g of pure alcohol) within 6 months before the first administration or who cannot abstain from consent to post-study visit.
* Heavy smoker (>10 cigarettes/day).

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Duration time with integrated gastric pH>4 / 24hr | 0-24hours

SECONDARY OUTCOMES:
Median 24 hr gastric pH | 0-24hours
Percent decrease from baseline in integrated gastric acidity for 24-hour interval after dose | 0-24hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk University Hospital, Cheongju-si, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Choi YS, Hwang JG, Kim JW, Min H, Seong CH, Hong SH, Kim NY, Park MK. Pharmacodynamics Between a Dual Delayed-Release Formulation of Low-Dose Esomeprazole and Famotidine in Healthy Korean Subjects. Clin Ther. 2024 Aug;46(8):622-628. doi: 10.1016/j.clinthera.2024.06.013. Epub 2024 Jul 20. PMID 39033046